CLINICAL TRIAL: NCT05275777
Title: A Phase Ib Safety lead-in, Followed by Phase II Trial of ADG106 in Combination With Neoadjuvant Doxorubicin and Cyclophosphamide Followed by Paclitaxel in Stage I-III HER2 Negative Breast Cancer
Brief Title: A Phase Ib Safety lead-in, Followed by Phase II Trial of ADG106 in Combination With Neoadjuvant Chemotherapy in HER2 Negative Breast Cancer
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National University Hospital, Singapore (Other)
Collaborators: Adagene Inc (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: ADG106-T6002
Record Dates: First submitted 2022-02-09; First posted 2022-03-11 (Actual); Last update posted 2025-07-25 (Actual); Status verified 2025-07

CONDITIONS: HER2-negative Breast Cancer; Advanced Solid Tumor
Keywords: HER2-negative Breast Cancer; ADG106; neoadjuvant doxorubicin and cyclophosphamide; paclitaxel
MeSH Terms: interventions — Doxorubicin; Cyclophosphamide; Paclitaxel

STUDY DESIGN:
Intervention Model Description: Phase Ib: A 3+3 dose escalation design will be used to determine the RP2D dose of ADG106 in combination with ddAC and paclitaxel respectively.
  Phase II: ADG106 will be combined with ddAC followed by paclitaxel as neoadjuvant chemotherapy in patients with stage I-III HER2 negative breast cancer.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- ADG106 combined with dose dense Doxorubicin and Cyclophosphamide (Phase Ib) (Experimental): Intravenous ADG106 + 2 weekly doxorubicin and cyclophosphamide
  Interventions: Drug: ADG106; Drug: Doxorubicin; Drug: Cyclophosphamide
- ADG106 combined with Paclitaxel (Phase Ib) (Experimental): Intravenous ADG106 + weekly paclitaxel
  Interventions: Drug: ADG106; Drug: Paclitaxel
- ADG106 combined with dose dense Doxorubicin and Cyclophosphamide follow by Paclitaxel (Phase II) (Experimental): Intravenous ADG106 combined with two weekly doxorubicin and cyclophosphamide followed intravenous ADG106 combined with weekly paclitaxel
  Interventions: Drug: ADG106; Drug: Doxorubicin; Drug: Cyclophosphamide; Drug: Paclitaxel

INTERVENTIONS:
Drug: ADG106 — Administered as an intravenous infusion over 60-90 minutes in the initial cycle and over 30 minutes in subsequent cycle if well tolerated.
Drug: Doxorubicin — Administered as an intravenous infusion.
  Other Names: Adriamycin
  Arms: ADG106 combined with dose dense Doxorubicin and Cyclophosphamide (Phase Ib); ADG106 combined with dose dense Doxorubicin and Cyclophosphamide follow by Paclitaxel (Phase II)
Drug: Cyclophosphamide — Administered as an intravenous infusion.
  Other Names: Cytophosphane
  Arms: ADG106 combined with dose dense Doxorubicin and Cyclophosphamide (Phase Ib); ADG106 combined with dose dense Doxorubicin and Cyclophosphamide follow by Paclitaxel (Phase II)
Drug: Paclitaxel — Administered as an intravenous infusion.
  Other Names: Taxol
  Arms: ADG106 combined with Paclitaxel (Phase Ib); ADG106 combined with dose dense Doxorubicin and Cyclophosphamide follow by Paclitaxel (Phase II)

SUMMARY:
This is an open label, lead in phase Ib dose confirmation study in patients with advanced solid tumors, followed by a phase II single arm study as neoadjuvant therapy in stage I-III HER2 negative breast cancer.

Primary Objectives

* To determine the safety profile of combination of ADG106 with dose dense doxorubicin/cyclophosphamide, and with weekly paclitaxel.
* To determine the Recommended Phase 2 Dose (RP2D) of ADG106 in combination with dose dense doxorubicin/cyclophosphamide, and with weekly paclitaxel.
* To evaluate biological changes on immunohistochemistry in HER2 negative breast cancer after treatment with ADG106 alone and in combination with chemotherapy.

Secondary Objectives

* To determine the efficacy of combination of ADG106 with standard neoadjuvant combination chemotherapy in HER2 negative breast cancer: objective response rates.
* To correlate tumor and plasma biomarkers with efficacy outcomes.

DETAILED DESCRIPTION:
The phase Ib segment will be carried out with a standard 3+3 dose de-escalation design. Patients with advanced/ metastatic solid organ cancers will be enrolled in 2 parallel cohorts.

Cohort 1 will receive ADG106 in combination with dose dense doxorubicin/ cyclophosphamide (AC).

Cohort 2 will receive ADG106 in combination with weekly paclitaxel.

In the phase II portion, patients with stage I-III HER2 negative breast cancer planned for neoadjuvant chemotherapy will be enrolled. Patients will be treated with neoadjuvant chemotherapy (ddAC followed by paclitaxel for 12 weeks) combined with ADG106, before definitive breast cancer surgery

ELIGIBILITY:
Inclusion Criteria:

Patients may be included in the study only if they meet all of the following criteria:

1. All patients must sign an informed consent in accordance with local institutional guidelines.
2. 18 years and above of age.
3. Estimated life expectancy of at least 12 weeks.
4. Has recovered from acute toxicities from prior anti-cancer therapies (phase Ib).
5. a) Phase Ib: Patients with histologically or cytologically confirmed advanced or metastatic solid tumors who have radiological evidence of progressive disease on study entry that are deemed likely to benefit from either dose dense doxorubicin/ cyclophosphamide or weekly paclitaxel.

   * There is no upper limit on the number of prior treatments provided all inclusion/ exclusion criteria are met. Hormone ablation therapy is considered an anti-cancer regimen. Radiation therapy and surgery are not considered anti-cancer regimens.
   * Prior receipt of immunotherapy is allowed. b) Phase II: Untreated stage I-III HER2 negative breast cancer patients who are planned for neoadjuvant chemotherapy followed by definitive breast cancer surgery.
6. Measurable disease by RECIST 1.1 criteria.
7. Eastern Cooperative Oncology Group (ECOG) Performance Status of 0-1.
8. Left ventricular ejection fraction of ≥ 50% for Cohort 1 in phase Ib and all patients in phase II.
9. Adequate bone marrow function and organ function within 2 weeks of study treatment.

   1. Adequate hematologic function defined as:

      * Absolute neutrophil count (ANC) ≥ 1.5 x 109/L
      * Platelets ≥ 100 x 109/L
      * Hemoglobin ≥ 9 x 109/L
   2. Adequate hepatic function defined as:

      * Bilirubin < 1.5 times the upper limit of normal (ULN)
      * ALT or AST < 2.5 times ULN (or < 5 times ULN with presence of liver metastases)
   3. Adequate renal function defined as:

      - Calculated creatinine clearance of ≥ 60 mL/min, calculated using the formula of Cockroft and Gault: (140-Age) x Mass (kg)/(72 x creatinine mg/dL); multiply by 0.85 if female.
   4. Adequate coagulation function defined as:

      * Activated partial thromboplastin time (aPTT) ≤1.5 x ULN
      * International normalized ratio (INR) ≤1.5 x ULN (Exception: INR 2 to ≤3 x ULN is acceptable for patients on warfarin anticoagulation
10. Patients with reproductive potential must use an approved contraceptive method if appropriate (e.g., intrauterine device, birth control pills, or barrier device) during and for three months after the study. Females with childbearing potential must have a negative serum pregnancy test within 7 days prior to study enrolment.
11. Able to comply with study related procedures.

Exclusion Criteria:

Patients will be excluded from the study for any of the following reasons:

1. Treatment within the last 30 days with any investigational drug.
2. Concurrent administration of any other tumor therapy, including cytotoxic chemotherapy, hormonal therapy, and immunotherapy.
3. Major surgery within 28 days of study drug administration.
4. Active infection that in the opinion of the investigator would compromise the patient's ability to tolerate therapy.
5. Serious concomitant disorders that would compromise the safety of the patient or compromise the patient's ability to complete the study, at the discretion of the investigator.
6. Active, known or suspected autoimmune disease. Subjects with type I diabetes mellitus, hypothyroidism only requiring hormone replacement, skin disorders (such as vitiligo, psoriasis, or alopecia) not requiring systemic treatment, or conditions not expected to recur in the absence of an external trigger are permitted to enrol.
7. Subjects with a condition requiring systemic treatment with either corticosteroids (>10mg daily prednisone equivalent) or other immunosuppressive medications within 14 days of randomization. Inhaled or topical steroids, and adrenal replacement steroid >10mg daily prednisone equivalent, are permitted in the absence of active autoimmune disease.
8. Subjects with interstitial lung disease that is symptomatic or may interfere with the detection or management of suspected drug-related pulmonary toxicity.
9. Known history of testing positive for human immunodeficiency virus (HIV) or known acquired immunodeficiency syndrome (AIDS).
10. Active hepatitis B (positive hepatitis B surface antigen [HBsAg]) or HCV (hepatitis C virus) [positive HCV RNA])

    1. Patients with past HBV infection or resolved HBV infection (defined as the presence of hepatitis B core antibody [HBcAb] and absence of HBsAg) are eligible. HBV DNA must be obtained in these patients prior to randomization. HBV carriers or those patients requiring antiviral therapy are not eligible to participate.
    2. Patients positive for HCV antibody are eligible only if PCR is negative for HCV RNA.
    3. HBV carriers or those subjects receiving antiviral treatment of hepatitis B virus or Hepatitis C are not eligible.
11. Pregnancy.
12. Breast feeding.
13. Second primary malignancy that is clinically detectable at the time of consideration for study enrolment. The exception is patients in phase II with two or more primary invasive breast cancers that are both HER2 negative and where both cancers are amenable to repeated biopsy. In this case, each tumor will be biopsied and assessed separately for treatment response.
14. Symptomatic brain metastases.
15. History of significant neurological or mental disorder, including seizures or dementia.
16. Unable to comply with study procedures.
17. Phase II cohort: Prior treatment for locally advanced or metastatic breast cancer.
18. Patients with known underlying hemoglobinopathies (e.g., thalassemia). Note: patients without known hemoglobinopathies do not specifically need to be screened for hemoglobinopathies in the absence of clinical suspicion).
19. History of life-threatening hypersensitivity or known to be allergic to protein drugs or recombinant proteins or any ingredients contained in the ADG106 drug formulation (succinic acid, arginine, polysorbate 80 and hydrochloric acid).
20. Peripheral neuropathy grade ≥2.
21. Live viral vaccine therapies within 4 weeks prior to the first dose of study drug.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Estimated)
Dates: Start 2022-05-19 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2030-02 (Estimated)

PRIMARY OUTCOMES:
Number of participant with treatment related toxicities | From enrolment till 30 days after last dose of study treatment
  Toxicities will be graded using the Common Terminology Criteria for Adverse Events (CTCAE) toxicity grading version 5.0.
Histological response after neoadjuvant ADG106 + chemotherapy | After 20 weeks of neoadjuvant chemotherapy
  Biological changes on immunohistochemistry will be evaluated using paraffin-embedded tumor specimens.

SECONDARY OUTCOMES:
Objective response rate in Phase Ib | At the end of every 3 cycles up to 24 weeks, at the end of every 6 cycles after 24 weeks up to 60 weeks (each cycle is 2 weeks)
  Complete and partial clinical response will be measured by RECIST 1.1.
Overall survival in Phase Ib | From enrolment till date of death or final follow up visit (maximum 1 year after last treatment dose)
  Defined as the time from the date of study enrolment to the date of death from any cause, regardless of whether the death occurred during the study or following treatment discontinuation.
Correlation of plasma biomarkers with efficacy outcome in Phase Ib | baseline, at the end of week 1, 2, 4, 6, 8, 10, 12, 14, 18, 30, 42, 54, 66
  Correlation of biomarkers with Objective Response Rate, Progression Free Survival, Overall Survival
Progression free survival in Phase Ib | From enrolment till disease progression or date of death or final follow-up visit (maximum 1 year after last treatment dose).
  Defined as the time from the date of study enrolment to the first date of documented disease progression.
Clinical response rate in Phase II | baseline, at the end of 2 weeks, 4 weeks, 8 weeks, 10 weeks, 12 weeks of treatment.
  Clinical response rate will be measured by calipers
Pathological complete response rate in Phase II | after 20 weeks neoadjuvant chemotherapy
  Defined as any patient who demonstrates no histological evidence of invasive tumor in the primary breast site as well as in resected axillary lymph nodes.
Relapse free survival in Phase II | From enrolment to final follow up visit (maximum 6 years from last treatment dose)
  Defined as the time from the date of study enrolment to the first date of documented disease relapse.

CONTACTS AND LOCATIONS:
Overall Officials: Soo Chin Lee, Principal Investigator — National University Hospital, Singapore
Locations (1):
- National University Hospital, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ding Y, Ding K, Yang H, He X, Mo W, Ding X. Does dose-dense neoadjuvant chemotherapy have clinically significant prognostic value in breast cancer?: A meta-analysis of 3,724 patients. PLoS One. 2020 May 29;15(5):e0234058. doi: 10.1371/journal.pone.0234058. eCollection 2020. PMID 32470093
- [Background] Hammerl D, Smid M, Timmermans AM, Sleijfer S, Martens JWM, Debets R. Breast cancer genomics and immuno-oncological markers to guide immune therapies. Semin Cancer Biol. 2018 Oct;52(Pt 2):178-188. doi: 10.1016/j.semcancer.2017.11.003. Epub 2017 Nov 6. PMID 29104025
- [Background] Nanda R, Liu MC, Yau C, Shatsky R, Pusztai L, Wallace A, Chien AJ, Forero-Torres A, Ellis E, Han H, Clark A, Albain K, Boughey JC, Jaskowiak NT, Elias A, Isaacs C, Kemmer K, Helsten T, Majure M, Stringer-Reasor E, Parker C, Lee MC, Haddad T, Cohen RN, Asare S, Wilson A, Hirst GL, Singhrao R, Steeg K, Asare A, Matthews JB, Berry S, Sanil A, Schwab R, Symmans WF, van 't Veer L, Yee D, DeMichele A, Hylton NM, Melisko M, Perlmutter J, Rugo HS, Berry DA, Esserman LJ. Effect of Pembrolizumab Plus Neoadjuvant Chemotherapy on Pathologic Complete Response in Women With Early-Stage Breast Cancer: An Analysis of the Ongoing Phase 2 Adaptively Randomized I-SPY2 Trial. JAMA Oncol. 2020 May 1;6(5):676-684. doi: 10.1001/jamaoncol.2019.6650. PMID 32053137
- [Background] Mittendorf EA, Zhang H, Barrios CH, Saji S, Jung KH, Hegg R, Koehler A, Sohn J, Iwata H, Telli ML, Ferrario C, Punie K, Penault-Llorca F, Patel S, Duc AN, Liste-Hermoso M, Maiya V, Molinero L, Chui SY, Harbeck N. Neoadjuvant atezolizumab in combination with sequential nab-paclitaxel and anthracycline-based chemotherapy versus placebo and chemotherapy in patients with early-stage triple-negative breast cancer (IMpassion031): a randomised, double-blind, phase 3 trial. Lancet. 2020 Oct 10;396(10257):1090-1100. doi: 10.1016/S0140-6736(20)31953-X. Epub 2020 Sep 20. PMID 32966830
- [Background] Schmid P, Cortes J, Pusztai L, McArthur H, Kummel S, Bergh J, Denkert C, Park YH, Hui R, Harbeck N, Takahashi M, Foukakis T, Fasching PA, Cardoso F, Untch M, Jia L, Karantza V, Zhao J, Aktan G, Dent R, O'Shaughnessy J; KEYNOTE-522 Investigators. Pembrolizumab for Early Triple-Negative Breast Cancer. N Engl J Med. 2020 Feb 27;382(9):810-821. doi: 10.1056/NEJMoa1910549. PMID 32101663
- [Background] Chu DT, Bac ND, Nguyen KH, Tien NLB, Thanh VV, Nga VT, Ngoc VTN, Anh Dao DT, Hoan LN, Hung NP, Trung Thu NT, Pham VH, Vu LN, Pham TAV, Thimiri Govinda Raj DB. An Update on Anti-CD137 Antibodies in Immunotherapies for Cancer. Int J Mol Sci. 2019 Apr 12;20(8):1822. doi: 10.3390/ijms20081822. PMID 31013788
- [Background] Ye L, Jia K, Wang L, Li W, Chen B, Liu Y, Wang H, Zhao S, He Y, Zhou C. CD137, an attractive candidate for the immunotherapy of lung cancer. Cancer Sci. 2020 May;111(5):1461-1467. doi: 10.1111/cas.14354. Epub 2020 Apr 3. PMID 32073704
- [Background] Makkouk A, Chester C, Kohrt HE. Rationale for anti-CD137 cancer immunotherapy. Eur J Cancer. 2016 Feb;54:112-119. doi: 10.1016/j.ejca.2015.09.026. Epub 2016 Jan 2. PMID 26751393
- [Background] Qian Y, Pei D, Cheng T, Wu C, Pu X, Chen X, Liu Y, Shen H, Zhang W, Shu Y. CD137 ligand-mediated reverse signaling inhibits proliferation and induces apoptosis in non-small cell lung cancer. Med Oncol. 2015 Mar;32(3):44. doi: 10.1007/s12032-015-0499-9. Epub 2015 Jan 29. PMID 25631633
- [Background] Brahmer JR, Lacchetti C, Schneider BJ, Atkins MB, Brassil KJ, Caterino JM, Chau I, Ernstoff MS, Gardner JM, Ginex P, Hallmeyer S, Holter Chakrabarty J, Leighl NB, Mammen JS, McDermott DF, Naing A, Nastoupil LJ, Phillips T, Porter LD, Puzanov I, Reichner CA, Santomasso BD, Seigel C, Spira A, Suarez-Almazor ME, Wang Y, Weber JS, Wolchok JD, Thompson JA; National Comprehensive Cancer Network. Management of Immune-Related Adverse Events in Patients Treated With Immune Checkpoint Inhibitor Therapy: American Society of Clinical Oncology Clinical Practice Guideline. J Clin Oncol. 2018 Jun 10;36(17):1714-1768. doi: 10.1200/JCO.2017.77.6385. Epub 2018 Feb 14. PMID 29442540